CLINICAL TRIAL: NCT06198309
Title: A Risk-predictive Model for Frequent Acute Exacerbation Phenotype in Patients With Severe Chronic Obstructive Pulmonary Disease
Brief Title: Risk Prediction Model for Exacerbating Phenotype in Patients With Chronic Obstructive Pulmonary Disease
Status: Recruiting | Type: Observational
Sponsor: Li An (Other)
Responsible Party: Sponsor-Investigator, Li An, chief physician, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Other Study IDs: al123456
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frequent exacerbation of COPD
- Non-frequent exacerbation of COPD

SUMMARY:
This study is planned to be conducted based on the cohort of patients with severe chronic obstructive pulmonary disease in our hospital. Based on gut microbiota, random forest was used to search for potential diagnostic biomarkers in patients with frequent acute exacerbation and controls with non frequent acute exacerbation; Construct a frequent acute exacerbation risk prediction model using random forest, support vector machine, and BP neural network models. The development of this study will provide valuable references for the clinical classification and prognosis evaluation of chronic obstructive pulmonary disease (COPD), and improve the health level of COPD patients by further searching for treatable targets.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria for COPD of the global initiative for chronic obstructive lung diseases (GOLD 2022) and GOLD grading Ⅲ - Ⅳ (FEV1/FVC<70%, FEV1% predicted value ≤ 50% after Bronchiectasis)
2. Age>40 years old
3. COPD stable for more than 4 weeks
4. Short acting Bronchiectasis was not used within 24 hours before this experiment, long acting Bronchiectasis was not used within 48 hours, and glucocorticoids were not used throughout the body in the past month
5. Patient informed and signed consent form

Exclusion Criteria:

1. Asthma, active pulmonary tuberculosis, interstitial pneumonia and severe Bronchiectasis
2. Complicated with serious diseases (acute infection, diabetes, stroke, heart disease, liver and kidney dysfunction, cancer or autoimmune disease)
3. History of chronic diarrhea or constipation
4. History of Gastrointestinal Surgery
5. Using probiotics or antibiotics within the past 4 weeks
6. No history of using oral hormones or traditional Chinese medicine in the past three months
7. Pregnancy or lactation

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A patient with severe chronic obstructive pulmonary disease who visited the Department of Respiratory and Critical Care Medicine, Beijing Chaoyang Hospital, Capital Medical University since January 2023
Sampling Method: Non-Probability Sample
Enrollment: 365 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the predictive performance of the COPD frequent seizure risk prediction model based on the area under the ROC curve. | A year
  According to the Area Under Curve (AUC) of ROC, the largest one has the best predictive performance. When AUC>0.5, the closer it is to 1, the better the predictive performance of the model. When AUC=0.5, it indicates poor model fitting and no potential predictive value.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China